CLINICAL TRIAL: NCT00463099
Title: Prognosis and Predictors of ACL Reconstruction - A Multicenter Cohort Study
Brief Title: Multicenter Orthopaedics Outcomes Network for ACL Reconstructions
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kurt P. Spindler, Adjoint Professor, Vanderbilt University Medical Center
Other Study IDs: 990426; R01AR053684 (NIH)
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Rupture of Anterior Cruciate Ligament
Keywords: Anterior Cruciate Ligament/injuries; Anterior Cruciate Ligament/surgery; Knee injuries/surgery; Outcomes research; Prospective Studies
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the effect of modifiable risk factors on knee function, osteoarthritis, and re-rupture of the anterior cruciate ligament (ACL) following ACL reconstruction.

DETAILED DESCRIPTION:
Disruption of the anterior cruciate ligament (ACL) is among the most frequent musculoskeletal injuries affecting physically active men and women. An estimated 200,000 ACL reconstructions (ACLR) are performed annually, and the incidence of this injury is roughly 1 in 3000 per year. ACL injury has both immediate and long-term implications for an injured person's quality of life, their risk for osteoarthritis (OA), and long-term disability. Currently, ACLR is recommended as the standard of care following an ACL tear based on evidence for improved instrumented laxity, the desire to return to sports play, and evidence for a reduction in future knee injuries.

In this research we propose to identify risk factors measurable at the time of injury/surgery in order to estimate the magnitude of the effect of these factors on important quality of life and clinical outcomes (e.g.,OA and incidence of additional surgery) 2 to 10 years after a patient's ACL reconstruction.

AIM 1. To identify risk factors for reduced quality of life 2-20 yrs post-ACLR, from information available at the time of surgery; including the characteristics of the patients (age, gender, body mass index, activity level, clinical knee alignment) and their injuries (concurrent meniscus, articular cartilage, and collateral ligament injuries), and treatment decisions made during the initial surgery (e.g., graft choice, meniscus and articular cartilage treatments).

AIM 2. To identify risk factors for symptoms and signs of osteoarthritis 2-20 years post-ACLR, from information available at the time of surgery; including the characteristics of the patients (as above) and their injuries (as above), and treatment decisions made during ACLR (as above).

AIM 3. To identify risk factors for recurrent ligament disruption and additional arthroscopic knee surgeries of the ACLR knee, from among the characteristics of the patients (as above), their initial injuries (as above), and treatment decisions made during ACLR (as above).

The overarching goal of this study is to establish evidence-based medicine practices of counseling patients on prognosis, guiding surgeons on treatment of meniscus and articular cartilage injuries, and post-surgical care, as well as the appropriate evidence for future interventional trials in the targeted subset of ACLRs with poorer outcomes.

ELIGIBILITY:
Inclusion Criteria:

- All ACL-deficient candidates scheduled for a unilateral ACL reconstruction at one of the participating MOON sites.

Exclusion Criteria:

* Persons undergoing a simultaneous bilateral ACL reconstruction
* Patients less than 10 years old and older than 80 years old
* Patients unwilling or unable to complete their follow-up questionnaire

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible ACL-deficient candidates scheduled for a unilateral ACL reconstruction at one of the participating MOON sites.
Sampling Method: Non-Probability Sample
Enrollment: 3294 (Actual)
Dates: Start 2002-01; Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
patient-reported outcome measures | 2, 6, 10, and 20 years
  Sports function (as measured by the KOOS and IKDC). Activity level (as measured by the Marx activity rating scale). General health (as measured by the SF-36).

SECONDARY OUTCOMES:
Signs and symptoms of osteoarthritis | 2, 6, 10, and 20 years
  Signs of OA (as measured by joint space narrowing on a standing radiograph). Symptoms of OA (as measured by WOMAC and KOOS pain subscales).

OTHER OUTCOMES:
ACL graft failure | 2, 6, 10, and 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Kurt P. Spindler, M.D., Principal Investigator — Vanderbilt University
Locations (8):
- United States (8):
  - University of Colorado, Boulder, Colorado
  - University of Iowa, Iowa City, Iowa
  - Washington University at St. Louis, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salem HS, Huston LJ, Zajichek A, McCarty EC, Vidal AF, Bravman JT, Spindler KP, Frank RM; MOON Knee Group; Amendola A, Andrish JT, Brophy RH, Jones MH, Kaeding CC, Marx RG, Matava MJ, Parker RD, Wolcott ML, Wolf BR, Wright RW. Anterior Cruciate Ligament Reconstruction With Concomitant Meniscal Repair: Is Graft Choice Predictive of Meniscal Repair Success? Orthop J Sports Med. 2021 Sep 14;9(9):23259671211033584. doi: 10.1177/23259671211033584. eCollection 2021 Sep. PMID 34541016
- [Derived] Marmura H, Getgood AMJ, Spindler KP, Kattan MW, Briskin I, Bryant DM. Validation of a Risk Calculator to Personalize Graft Choice and Reduce Rupture Rates for Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2021 Jun;49(7):1777-1785. doi: 10.1177/03635465211010798. Epub 2021 May 4. PMID 33945339